CLINICAL TRIAL: NCT06963463
Title: Transdiagnostic Sleep and Circadian Intervention + Bright Light in Adolescents With Elevated Depression
Brief Title: Transdiagnostic Sleep and Circadian Intervention + Bright Light in Adolescents With Elevated Depression (TranS-C+BL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Oregon (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tina R Goldstein, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22040040; P50MH115838 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disturbance; Sleep; Depression; Suicide
Keywords: Sleep Disturbances; Objective Sleep; Subjective Sleep Difficulties; Minority Youth
MeSH Terms: conditions — Parasomnias; Depression; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Feedback (Experimental): Participants receive an actigraphy watch to track their sleep and activity levels and complete a daily sleep diary; sleep feedback graphs show participants their actigraphy watch and sleep diary data on demand.
  Interventions: Behavioral: Sleep Feedback
- TranS-C + Sleep Feedback (Experimental): Participants will attend 6-8 TranS-C sessions with a Sleep therapist. Participants will also wear bright light glasses in the morning and blue light blocking glasses in the evening throughout the intervention.
  Interventions: Behavioral: TranS-C; Behavioral: Sleep Feedback

INTERVENTIONS:
Behavioral: TranS-C — This intervention includes participants attending 6-8 sessions with a Sleep Therapist.
  Arms: TranS-C + Sleep Feedback
Behavioral: Sleep Feedback — Participants are provided with an actigraphy watch that is used to monitor their sleep and activity throughout the day and complete a sleep diary daily. Along with wearing the watch they also will be provided access to their actigraphy and sleep diary graphs that document their data.

SUMMARY:
The goal of this clinical trial is to adapt a sleep intervention for individuals representative of all demographic groups, including those who are at the highest risk for suicidal behavior. Sleep difficulties are a promising target for youth with suicidal thoughts and behavior to focus on as a prevention measure. We aim to increase intervention acceptability and impact by adapting it for the adolescent populations at highest risk for suicidal thoughts and behavior. The research project will compare Transdiagnostic Sleep and Circadian Intervention (TranS-C), an evidence based, modularized intervention that targets a range of sleep difficulties to a treatment as usual or control condition including providing weekly sleep feedback reports from data entered into a daily sleep diary and from wearing a sleep sensing, actigraphy watch. Participants in both conditions (TranS-C vs. Sleep Feedback) will wear an actigraphy sleep watch that monitors sleep, and complete daily sleep diaries via smartphone or email. Participants in the TranS-C condition will also wear bright light (BL) and blue blocking glasses each day as well as attend weekly or biweekly sessions with a Sleep Therapist. The sleep therapist will review sleep feedback during sessions.

DETAILED DESCRIPTION:
This study will adapt TranS-C+BL for at-risk adolescents using health equity-informed implementation science methods.

This randomized trial will enroll 75 youth aged 12-18 at risk for STB and clinically significant sleep difficulties identified in primary care. The randomization that this study uses is a 2:1 allocation to compare TranS-C+BL Sleep Feedback vs. Sleep Feedback Alone.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (12-18)
* Current moderate to severe depression as measured by the PHQ-9M with a total score of greater than or equal to 11
* Current clinically significant sleep disturbance measured by the PHQ-9-M sleep item greater than or equal to 2.
* English language fluency and literacy sufficient to engage in study protocol.

Exclusion Criteria:

* Evidence of obstructive sleep apnea,
* Evidence of restless legs syndrome
* Evidence of psychosis
* Evidence of bipolar disorder
* Evidence of a developmental disability precluding comprehension of study procedures per electronic health record and eligibility screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility-Attendance | From enrollment to the end of the treatment (up to 4 months)
  Feasibility of interventions as by measured by the mean of number of sessions attended. Local study documents are used to track each session that was completed.
Feasibility-Attrition | From enrollment until withdrawal or completing treatment sessions.
  Attrition will be assessed using a study-specific form reflecting participants who withdraw or are withdrawn from the TranS-C+ intervention. The proportion of patients who withdraw or are withdrawn will be calculated.
Acceptability-Treatment Satisfaction | 4 month
  Treatment satisfaction will be measured by the patient-reported Treatment Satisfaction Questionnaire administered post-treatment. The Treatment Satisfaction Questionnaire assesses satisfaction with the treatment received and perception of progress; each item is rated on a Likert scale. Additional open-ended questions allow for participants to share feedback on strengths and weaknesses as well as any other feedback related to their satisfaction with the intervention. The Questionnaire has questions on a 1(Not at all)-7(Very Much). Questions on study clinicians are asked on a 1(Poor)-7(Superior) Likert scale. Questions on the duration of study on a 1(Much too short)-7(Much to long) Likert scale. Questions about frequency of visits on a 1(Much too infrequent)-7(Much to frequent). Questions for recommendations to other rated on a 1(Strongly recommend)-7(Strongly not recommend). Questions on future outlook rated on a 1(Very Pessimistic)-7(Very Optimistic).

SECONDARY OUTCOMES:
Sleep Disturbance | Baseline
  Self-reported sleep disturbance will be assessed via the Pediatric PROMIS Sleep Disturbance and Sleep Related Impairment Measures. The Patient-Reported Outcomes Measurement Information System is an 8-item measure. The scoring ranges from Never (1) Almost Never (2) Sometimes (3) Almost Always (4) Always (5). The PROMIS scale is scored on the T-score metric scale. The higher the participant scores more of the concept being measured. With the general population getting a score of 50 with a standard deviation of 10
Depression | Baseline
  Depressive symptom severity will be assessed via the self-reported PHQ-9-M. The Patient Health Questionnaire is a 13-item measure. The questions are rating on a 0(Not at all)- 3(Nearly Every day) Likert scale. Additional questions rated on a scale of Not difficult at all to Extremely difficult, along with yes/no questions. The PHQ-9M is rated on a scale from 0 to 27. Higher scores are associated with higher levels of, or more severe, depression
Risk for Suicidal Thoughts and Behaviors | Baseline
  Suicidal thoughts and behaviors will be assessed via the C-SSRS. The Columbia-Suicide Severity Rating Scale is an 18-item measure. This measure contains yes/no questions, asking about both about suicidality over the past 3 months and lifetime. In the C-SSRS the higher the score the more risk of suicidality (0 = No risk reported (all "no" responses),1 - 2 = Low risk ,3 - 6 = Moderate to high risk)
Sleep Disturbance | 1 month
  Self-reported sleep disturbance will be assessed via the Pediatric PROMIS Sleep Disturbance and Sleep Related Impairment Measures. The Patient-Reported Outcomes Measurement Information System is an 8-item measure. The scoring ranges from Never (1) Almost Never (2) Sometimes (3) Almost Always (4) Always (5). The PROMIS scale is scored on the T-score metric scale. The higher the participant scores more of the concept being measured. With the general population getting a score of 50 with a standard deviation of 10
Sleep Disturbance | 4 months
  Self-reported sleep disturbance will be assessed via the Pediatric PROMIS Sleep Disturbance and Sleep Related Impairment Measures. The Patient-Reported Outcomes Measurement Information System is an 8-item measure. The scoring ranges from Never (1) Almost Never (2) Sometimes (3) Almost Always (4) Always (5). The PROMIS scale is scored on the T-score metric scale. The higher the participant scores more of the concept being measured. With the general population getting a score of 50 with a standard deviation of 10
Depression | 1 month
  Depressive symptom severity will be assessed via the self-reported PHQ-9-M. The Patient Health Questionnaire is a 13-item measure. The questions are rating on a 0(Not at all)- 3(Nearly Every day) Likert scale. Additional questions rated on a scale of Not difficult at all to Extremely difficult, along with yes/no questions. The PHQ-9M is rated on a scale from 0 to 27. Higher scores are associated with higher levels of, or more severe, depression
Depression | 4 month
  Depressive symptom severity will be assessed via the self-reported PHQ-9-M. The Patient Health Questionnaire is a 13-item measure. The questions are rating on a 0(Not at all)- 3(Nearly Every day) Likert scale. Additional questions rated on a scale of Not difficult at all to Extremely difficult, along with yes/no questions. The PHQ-9M is rated on a scale from 0 to 27. Higher scores are associated with higher levels of, or more severe, depression
Risk for Suicidal Thoughts and Behaviors | 1 month
  Suicidal thoughts and behaviors will be assessed via the C-SSRS. The Columbia-Suicide Severity Rating Scale is an 18-item measure. This measure contains yes/no questions, asking about both about suicidality over the past 3 months and lifetime. In the C-SSRS the higher the score the more risk of suicidality (0 = No risk reported (all "no" responses),1 - 2 = Low risk ,3 - 6 = Moderate to high risk)
Risk for Suicidal Thoughts and Behaviors | 4 month
  Suicidal thoughts and behaviors will be assessed via the C-SSRS. The Columbia-Suicide Severity Rating Scale is an 18-item measure. This measure contains yes/no questions, asking about both about suicidality over the past 3 months and lifetime. In the C-SSRS the higher the score the more risk of suicidality (0 = No risk reported (all "no" responses),1 - 2 = Low risk ,3 - 6 = Moderate to high risk)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Goldstein, Ph.D, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the NIMH's data sharing and data use policies this research study and clinical trial will be compliant with requirements for depositing data with the NIMH Data Archive (NDA) in the National Database for Clinical Trials Related to Mental Illness (NDCT). Specific statements will be added to the consent forms to allow for data sharing. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies.
Time Frame: Individual participant data will be available in a deidentified manner through the NIMH Data Archive indefinitely.
Access Criteria: Verified researchers may request the data through the NIMH Data Archive.